CLINICAL TRIAL: NCT00947830
Title: A Study Investigating the Predictive Value of Intracellular and Plasma Imatinib Levels in Newly Diagnosed Patients With Chronic Myeloid Leukemia
Brief Title: Investigating Intracellular and Plasma Imatinib Levels in Chronic Myeloid Leukemia
Acronym: OCT-1
Status: Completed | Type: Observational
Sponsor: Brian Leber (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor-Investigator, Brian Leber, Professor of Medicine, Hamilton Health Sciences Corporation
Organization: McMaster University (Other)
Other Study IDs: OCT-1
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; intracellular imatinib level; OCT-1
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood cells
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to find out if the level of imatinib in the bloodstream, and the level that leukemia cells will predict how quickly your chronic myeloid leukemia improves with the treatment.

1.1 Primary Objectives

To determine if intracellular levels of Imatinib in leukemic blood cells within two weeks of treatment initiation of patients with chronic myeloid leukemia in chronic phase predicts molecular and cytogenetic response at 6 and 12 months post treatment

1.2. Secondary Objectives

1.2.1 To determine if hOCT-1 mRNA levels at diagnosis predict Imatinib intracellular levels within two weeks of treatment initiation.

1.2.2 To determine the correlation between intracellular Imatinib levels at two weeks of treatment initiation with plasma Imatinib levels at two and four weeks after treatment initiation.

1.2.3 To determine if plasma Imatinib levels four weeks after treatment initiation correlate with plasma Imatinib levels 12 months after treatment initiation.

1.2.4 To determine if intracellular levels of Imatinib in leukemic blood cells within two weeks of treatment initiation correlate with intracellular levels of Imatinib in normal leukocytes 12 months after treatment initiation.

DETAILED DESCRIPTION:
The use of imatinib for the treatment of chronic myeloid leukemia has significantly improved the survival of most patients with this disease. This drug works by directly inhibiting the cancer-causing protein BCR-ABL that is found inside the leukemia cells and therefore is the first successful targeted treatment for cancer. Measuring the amount of the gene product for BCR-ABL by very sensitive laboratory techniques as it decreases during therapy has been extremely helpful in monitoring disease activity. Furthermore, in a subgroup of patients whose leukemia cells decrease by more than a thousand-fold measured by this sensitive technique during the first one or two years, these patients have a greater than 97% chance that disease remains under excellent control for more than five years. Therefore, discovering tests that would predict this marked decrease in BCR-ABL gene product at early timepoints when any treatment changes could be done would be very useful. To study this, a test that measures the amount of imatinib in a patient's bloodstream plasma has been recently developed at a national reference laboratory, Warnex Medical Laboratories in Laval, Quebec. Preliminary results from other national laboratories indicates that patients differ in how much imatinib their bodies absorb and get into their bloodstream, and that patients who absorb imatinib less well have a slightly lower chance of this thousand-fold reduction in leukemia levels. However, because imatinib must get inside leukemia cells to inhibit BCR-ABL, it likely that the amount of imatinib that is inside leukemia cells would predict even better the response to the drug. Warnex Laboratories has recently developed a test that can measure imatinib levels inside cells, and preliminary results indicate that patients differ in how much imatinib gets inside their cells. Dr. Suzanne Kamel-Reid's laboratory at Toronto General Hospital has also developed a test to measure the amount of gene product for the pore that imatinib uses to enter leukemia and other blood cells (called h-OCT-1), and her preliminary results also show that differs among patients. It is not clear if these differences are due to differences in the leukemia cels themselves between patients, or in differences between the way imatinib would get into any blood cells between patients. Therefore we are undertaking this current study to see (1) which of the tests, or combination of tests (bloodstream imatinib level, imatinib level inside cells, or h-OCT-1 level) best predicts how well patients patients respond to imatinib by the sensitive test for BCR-ABL, and (2) whether the differences between patients in the level inside cells is due specifically to the leukemia cells. In this trial, we will measure these levels on patients who are about to begin treatment for their chronic myeloid leukemia with imatinib. For practical purposes, participation in this trial would require patients to have extra blood samples drawn at several visits when they would normally see their hematologist/oncologist to monitor their disease and its treatment: within 28 days up to and including Day 1 as long as collected prior to start of treatment with Imatinib, and once Imatinib treatment is started, at 2 weeks, one month, 6 months , and 12 months. By obtaining this information, we may better understand how to adjust imatinib therapy to achieve the best response for more patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of chronic myeloid leukemia in chronic phase (as defined in Appendix A) within four weeks of study registration based on bone marrow aspirate and peripheral blood counts. - Patients must have confirmation of the Philadelphia chromosome or variants by cytogenetics, or FISH, or positive test for bcr-abl by PCR. Patients with additional chromosomal abnormalities in addition to the Philadelphia chromosome are eligible.
* Age >18 years.
* ECOG performance status <2. (Appendix B)
* Patients must have normal organ function as defined below:

  * Total Bilirubin < 1.5 x Institutional Upper Limit of Normal (ULN)
  * AST and/or ALT < 2.5 x Institutional Upper Limit of Normal (ULN)
* Eligibility of patients receiving any medications or substances known to affect or determined following review of their case by the Principal Investigator.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents.
* Patients may not have received prior treatment with Imatinib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women are excluded from this study because Imatinib has potential teratogenic effects and excretion in breast milk is unknown.
* No prior malignancies except for: adequately treated non-melanoma skin cancer, cervical carcinoma-in-situ, adequately treated Stage I or II cancer from which patient is in complete remission, or any other cancer from which patient has been disease free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed patients with chronic myeloid leukemia in chronic phase
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To determine if intracellular levels of Imatinib in leukemic blood cells within two weeks of treatment initiation of patients with chronic myeloid leukemia in chronic phase predicts molecular and cytogenetic response at 6 and 12 months post treatment | One year after starting therapy for chronic myeloid leukemia

SECONDARY OUTCOMES:
To determine if hOCT-1 mRNA levels at diagnosis predict Imatinib intracellular levels, OCT-1 levels at one year | One year after starting therapy for chronic myeloid leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leber, MDCM, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada